CLINICAL TRIAL: NCT04230772
Title: A Randomized Controlled Trial Comparing Clinical Outcomes of Natural Orifice Specimen Extraction Surgery Versus Traditional Robotic-assisted Surgery for Patients With Colorectal Cancer
Brief Title: Clinical Outcomes of NOSES Versus Traditional Robotic-assisted Surgery for Patients With Colorectal Cancer
Acronym: NOTR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taiyuan Li (Other)
Responsible Party: Sponsor-Investigator, Taiyuan Li, Prof., Chief physician, Head of The Fifth Department of General Surgery, The First Affiliated Hospital of Nanchang University
Organization: The First Affiliated Hospital of Nanchang University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ndyfy660618
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Colorectal Neoplasms; Neoplasms Malignant; Complication of Surgical Procedure; Robotic Surgical Procedures; Natural Orifice Specimen Extraction Surgery
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Natural Orifice Specimen Extraction Surgery (Experimental): Natural orifice specimen extraction surgery will performed in patients assigned to this group.
  Interventions: Procedure: Natural Orifice Specimen Extraction Surgery
- Traditional Robotic-assisted Surgery (Active Comparator): Traditional robotic-assisted surgery will performed in patients assigned to this group.
  Interventions: Procedure: Traditional Robotic-assisted Surgery

INTERVENTIONS:
Procedure: Natural Orifice Specimen Extraction Surgery — In the experimental group, patients will be performed robotic colorectal resection with natural orifice specimen extraction.
  Arms: Natural Orifice Specimen Extraction Surgery
Procedure: Traditional Robotic-assisted Surgery — In the active comparator group, patients will be performed traditional robotic-assisted colorectal resection.
  Arms: Traditional Robotic-assisted Surgery

SUMMARY:
In this study, the investigators will compare the clinical outcomes of the natural orifice specimen extraction surgery versus traditional robotic-assisted surgery in the treatment of colorectal cancer.

DETAILED DESCRIPTION:
Based on investigators' experience, compared to robotic-assisted colorectal cancer radical resection, robotic colorectal cancer radical resection with natural orifice extraction has more advantages in postoperative stress response, postoperative pain, postoperative recovery and postoperative abdominal aesthetics. However, in terms of tumor radicality, there may be no obvious differences. There are no randomized controlled trails to discuss these questions.This research is based on the above conditions. Investigators use prospective randomized controlled trial to analyze the surgical data, postoperative complications, postoperative recovery of the robotic colorectal cancer radical resection with natural orifice extraction and conventional robotic-assisted colorectal cancer radical resection in order to summarize clinical experience and explore the advantages and disadvantages of robotic colorectal cancer radical resection with natural orifice specimen extraction and to provide a new direction for the surgical treatment of colorectal cancer, which is beneficial to the promotion of NOSES(Natural Orifice Specimen Extraction Surgery ) technology and treatment of colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 80 years;
2. Performance status of 0 or 1 on ECOG (Eastern Cooperative Oncology Group) scale;
3. Histological or cytological confirmation of colorectal adenocarcinoma;
4. High rectal and sigmoid cancer with the lower margin of the tumor greater than 10 cm from the anal dentate line;
5. T1-3N0M0 at preoperative evaluation according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual 8th Edition, Transvaginal NOSES procedure w specimen with a circumferential diameter of <5 cm;
6. Preoperative examination did not suggest distant metastasis, implantation or invasion of adjacent organs;
7. Cardiopulmonary liver and kidney function can withstand surgery;
8. Written informed consent for participation in the trial.

Exclusion Criteria:

1. Not suitable for robot laparoscopic surgery;
2. The tumor is too large to be pulled out through the anus or vagina;
3. Simultaneous multiple primary cancer;
4. Emergency surgery due to complication (bleeding, obstruction or perforation) caused by primary cancer
5. Women with acute gynecological infections, vaginal deformities, unmarried and infertile women and women who are married and plan to get pregnant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of surgical complications | 30 days
  Complication rate of surgery within 30 days after surgery.

SECONDARY OUTCOMES:
The variation of C-reactive protein | Preoperative 3 days and postoperative 1, 3, and 7 days
  The values of C-reactive protein from peripheral blood before operation and on postoperative day 1, 3, 7 are recorded to access the surgical response stress and immune response.
The variation of interleukin-6(IL-6) | Preoperative 3 days and postoperative 1, 3, and 7 days
  The values of interleukin-6(IL-6) from peripheral blood before operation and on postoperative day 1, 3, 7 are recorded to access the surgical response stress and immune response.
The variation of interleukin-10(IL-10) | Preoperative 3 days and postoperative 1, 3, and 7 days
  The values of interleukin-10(IL-10) from peripheral blood before operation and on postoperative day 1, 3, 7 are recorded to access the surgical response stress and immune response.
The variation of cortisol | Preoperative 3 days and postoperative 1, 3, and 7 days
  The values of cortisol from peripheral blood before operation and on postoperative day 1, 3, 7 are recorded to access the surgical response stress and immune response.
The variation of lymphocyte subsets count of CD3, CD4 and CD8 | Preoperative 3 days and postoperative 1, 3, and 7 days
  The values of lymphocyte subsets count of CD3, CD4 and CD8 from peripheral blood before operation and on postoperative day 1, 3, 7 are recorded to access the surgical response stress and immune response.
The positive rate of malignant cells in ascitic fluid specimen | 1 day
  Ascitic fluid specimen will be taken after surgery and tested by clinical laboratory.
The positive rate of bacterial culture in ascitic fluid specimen | 1 day
  Ascitic fluid specimen will be taken after surgery and tested by clinical laboratory.
Postoperative pain score | 1 day
  Postoperative pain score will be assessed by visual analog score.
Time to first flatus | 30 days
  Time to first flatus is used to assess the postoperative recovery course
Time to leave bed postoperatively | 30 days
  Time to first leave bed postoperatively in hours is used to assess the postoperative recovery course.
Time to first liquid diet postoperatively | 30 days
  Time to first liquid diet postoperatively in days is used to assess the postoperative recovery course.
Postoperative hospital stay | 30 days
  Postoperative hospital stay is used to assess the postoperative recovery course.
Operation time | 1 day
  Time from start of incision to finish of abdominal closure.
Estimated blood loss | 1 day
  Blood loss will be measured according to the suction and the weight of wet gauze, and then minus the irrigation.
Number of retrieved lymph nodes | 1 day
  Number of retrieved lymph nodes will be determined according to the pathological report.

CONTACTS AND LOCATIONS:
Overall Officials: Taiyuan Li, M.D., Ph.D, Principal Investigator — Department of General Surgery, The First Affiliated Hospital of Nanchang University
Locations (7):
- China (7):
  - Chinese PLA General Hospital (301 Hospital) China, Beijing, Beijing Municipality
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - First Affiliated Hospital of Gannan Medical College, Ganzhou, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luo R, Zheng F, Zhang H, Zhu W, He P, Liu D. Robotic natural orifice specimen extraction surgery versus traditional robotic-assisted surgery (NOTR) for patients with colorectal cancer: a study protocol for a randomized controlled trial. Trials. 2021 Feb 6;22(1):121. doi: 10.1186/s13063-021-05077-z. PMID 33549133